CLINICAL TRIAL: NCT04333056
Title: Comparison of Two Swept-Source Optical Coherence Tomography-based Biometry Devices
Brief Title: Comparison Between Two Ss-OCT Biometry
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Ophthalmology Department, principal investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: ss-OCT biometry comparison
Record Dates: First submitted 2020-03-28; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Cataract Senile
Keywords: biometry; ss-OCT; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biometric measurement agreement — Patients scheduled for cataract surgery were measured with both ss-OCT devices. The following biometry parameters were compared: anterior keratometry, central corneal thickness (CCT), anterior chamber depth (ACD), lens thickness (LT) and axial length (AL).

SUMMARY:
Since recently a second swept-source optical coherence tomography (ss-OCT) optical biometry device was launched (Anterion, Heidelberg Engineering). Aim of this study is a retrospective data collection of patients who were measured with both ss-OCT optical biometry devices and to assess the limits of agreement of the two devices.

Retrospective comparison of two ss-OCT biometry devices concerning comparability of measurements of axial eye length, anterior chamber depth, lens thickness and keratometry.

DETAILED DESCRIPTION:
This a retrospective study including data acquired from patients that attended pre-surgical examination as it is the standard in the investigator's hospital.

The IOL Master 700 (Carl Zeiss Meditec AG, Jena) and the Heidelberg Anterion (Heidelberg Engineering, Germany) are biometry devices that use swept-source optical coherence tomography technology in combination with a multidot-keratometer, that obtain two-dimensional images of ocular structures.

The difference between the two devices resides in the wavelength of the infrared laser: 1200-1400nm for the Anterion and 1050nm for the IOL Master 700.

The SS-OCT devices provide a scan depth of 44mm and a resolution in tissue of 22 μm for the IOL Master 700 and of 14x16.5 mm and 30 μm for the Heidelberg Anterion.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract

Exclusion Criteria:

* nystagmus
* physical inabilities that could interfere with fixation
* dens cataract
* macular or corneal pathologies that could compromise fixation during the measurements.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were selected by the clinical investigators at the Hanusch Hospital.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Limits of agreement between two optical biometers using the same SS-OCT technology for the following parameters AL, ACD, LT (evaluated in mm) | 6 months
  For descriptive analysis, Kolmogorov Smirnov test will be used to evaluate normal distribution.
  The student T test for paired samples and Wilcoxon for nonparametric data was used to compare parameters as: AL, ACD, LT.
  The limits of agreement (1.96xSD) between two optical biometers were calculated and represented graphically using Bland-Altman graphs
Limits of agreement between two optical biometers using the same SS-OCT technology for the following parameters CCT (evaluated in micrometer) | 6 months
  For descriptive analysis, Kolmogorov Smirnov test will be used to evaluate normal distribution.
  The student T test for paired samples and Wilcoxon for nonparametric data was used to compare the CCT data The limits of agreement (1.96xSD) between two optical biometers were calculated and represented graphically using Bland-Altman graphs
Limits of agreement between two optical biometers using the same SS-OCT technology for the following parameter: keratometry (evaluated in diopter) | 6 months
  For descriptive analysis, Kolmogorov Smirnov test will be used to evaluate normal distribution.
  The student T test for paired samples and Wilcoxon for nonparametric data was used to compare keratometry data The limits of agreement (1.96xSD) between two optical biometers were calculated and represented graphically using Bland-Altman graphs

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., MD, Principal Investigator — VIROS, Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisus AD, Hirnschall ND, Findl O. Comparison of 2 swept-source optical coherence tomography-based biometry devices. J Cataract Refract Surg. 2021 Jan 1;47(1):87-92. doi: 10.1097/j.jcrs.0000000000000373. PMID 32769752